CLINICAL TRIAL: NCT06696430
Title: Nudging (Influencing Behavior and Decisions) to Promote the Use of Transcutaneous Electrical Nerve Stimulation for Postoperative Pain Relief
Brief Title: Nudging to Promote the Use of Transcutaneous Electrical Nerve Stimulation for Postoperative Pain Relief
Acronym: Nudging pain
Status: Recruiting | Type: Observational
Sponsor: Pether Jildenstal (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Pether Jildenstal, Professor, PhD, Göteborg University
Organization: Göteborg University (Other)
Other Study IDs: 2024-06961-01; 2024-06961-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2024-11-13; First posted 2024-11-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Postoperative Pain in Urological Surgery; Pain Management in Postoperative Care (Including Opioid-Sparing Approaches)
Keywords: Transcutaneous Electrical Nerve Stimulation (TENS); Nudging; Multimodal Analgesia; Postoperative Pain Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group (Baseline): This group includes healthcare staff and patients prior to the intervention. Baseline data will be collected on TENS usage rates, pain levels, and opioid consumption to assess initial practices in postoperative pain management.
- Intervention Group X1 (Education + superusers): Healthcare staff and patients following an educational intervention. This phase includes sessions on TENS usage and support from designated "superusers" to increase knowledge and skills related to TENS for postoperative pain management.
  Interventions: Behavioral: Educational Intervention on TENS Usage
- Intervention Group X2 (Nudging): Healthcare staff exposed to nudging strategies designed to enhance the use of TENS, which is currently available in routine care but underutilized. This phase involves visual prompts, reminders, and environmental cues aimed at making TENS more salient and encouraging its use for postoperative pain management.
  Interventions: Behavioral: Nudging Intervention to Promote TENS Usage

INTERVENTIONS:
Behavioral: Educational Intervention on TENS Usage — Educational sessions on TENS usage and support from designated "superusers" to increase knowledge and skills related to TENS for postoperative pain management.
  Groups: Intervention Group X1 (Education + superusers)
Behavioral: Nudging Intervention to Promote TENS Usage — Healthcare staff exposed to nudging strategies designed to enhance the use of TENS, which involves visual prompts, reminders, and environmental cues aimed at making TENS more salient and encouraging its use for postoperative pain management.
  Groups: Intervention Group X2 (Nudging)

SUMMARY:
This study aims to increase the use of transcutaneous electrical nerve stimulation (TENS) for acute postoperative pain relief. TENS, a non-pharmacological treatment using electrical impulses, can enhance pain relief, reduce opioid use, and minimize side effects. Despite its benefits, TENS is underused in healthcare. This project will provide TENS education, support from experienced "superusers," and nudging techniques to encourage staff to adopt TENS, ultimately improving pain management and recovery for postoperative patients.

DETAILED DESCRIPTION:
This research project investigates the effectiveness of combining educational initiatives, support from designated "superusers," and behavioral nudging to enhance the use of transcutaneous electrical nerve stimulation (TENS) in postoperative pain management. TENS, a non-pharmacological treatment, has shown effectiveness in alleviating postoperative pain, reducing opioid requirements, and improving patient recovery. Despite these benefits, TENS remains underutilized due to knowledge gaps, cultural, and organizational barriers. This project will explore how targeted interventions can drive TENS adoption, aiming to position it as an integral part of multimodal analgesia for postoperative care.

Outcomes

The study targets both staff and patient outcomes. Expected outcomes include:

* Primary Outcomes: Increased frequency of TENS usage among healthcare staff for postoperative pain, patient-reported reduction in pain intensity, and shortened discharge times.
* Secondary Outcomes: Reduced reliance on opioid pain relief, improved patient-reported postoperative experience (e.g., pain relief, symptom control for urinary urgency and bladder spasms), and healthcare staff's perceptions of nudging and educational interventions.

Methods

The project consists of three studies:

1. Quasi-Experimental Study (Study I):

   * Design: A pretest-posttest design with three observation periods (baseline, post-education, and post-nudging intervention).
   * Intervention: Staff receive TENS training through workshops, instructional videos, and hands-on support from "superusers" trained in TENS administration. Following the educational phase, nudging techniques (e.g., visual reminders, posters) are introduced to promote TENS as a default option for postoperative pain.
   * Data Collection: Baseline and follow-up data collection on TENS usage rates, patient demographics, pain intensity (using Visual Analog Scale/Numerical Rating Scale), opioid consumption, and discharge times.
2. Healthcare Staff Interviews (Study II):

   * Design: Qualitative interviews with 20-25 anesthesia staff members.
   * Focus: Describing anesthesia staff experiences with the nudging and educational interventions, perceived barriers to TENS adoption, and attitudes towards non-pharmacological pain management.
   * Data Collection: In-depth thematic analysis of interview responses to identify factors influencing TENS usage and the effectiveness of behavioral nudges.
3. Patient Interviews (Study III):

   * Design: Qualitative interviews with 20-25 patients who underwent robotic prostate surgery and received TENS for pain management.
   * Focus: Investigating patient experiences with TENS in managing pain and postoperative symptoms, particularly urinary urgency and bladder spasms.
   * Data Collection: Interviews conducted within one day post-discharge to capture immediate impressions of TENS's impact on pain relief and recovery quality.

Data Collection and Analysis

Data will be collected across approximately 500 patients in Study I and through thematic interviews with staff and patients in Studies II and III. Statistical analyses will include:

* Descriptive Statistics: To assess TENS usage frequency and patient-reported pain levels.
* T-Tests and Chi-Square Tests: For comparing pre- and post-intervention TENS adoption rates and categorical data.
* ANOVA and Multivariate Regression: To evaluate differences across intervention phases and control for confounding factors.
* Qualitative Thematic Analysis: Applied to staff and patient interview data to extract themes related to TENS acceptance, nudging impact, and the perceived effectiveness of educational interventions.

ELIGIBILITY:
Inclusion Criteria:

* All staff working in the department where the study will be conducted.
* Patients scheduled for urological procedures under anesthesia who are 18 years of age or older.

Exclusion Criteria:

* Does not give consent.
* Ongoing pregnancy.
* Unable to speak or understand Swedish.
* Presence of electronic implants (e.g., pacemaker, implantable - defibrillator/ICD).
* Regular preoperative use of opioids.
* Chronic pain condition.
* Known substance abuse.
* Reduced sensation at the site for TENS application.
* Severe untreated psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes healthcare staff working in the department where the study is conducted and patients who are scheduled for urological procedures under anesthesia and are 18 years or older. The focus is on observing and enhancing TENS usage in postoperative pain management within this specific clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of TENS Usage in Postoperative Care | 12 weeks (over the course of the intervention phases)
  Measure the frequency and consistency of TENS usage by healthcare staff for postoperative pain management across the three groups (Control, Education, and Nudging). This outcome will determine the effectiveness of educational and nudging interventions in changing TENS adoption patterns. Scores represent the number of documented TENS applications per patient.

SECONDARY OUTCOMES:
Change in Postoperative Pain Intensity | 1 day post-surgery, measured during patient recovery
  Assess patient-reported pain intensity using the Visual Analog Scale (VAS) or Numerical Rating Scale (NRS) to evaluate the impact of TENS on pain relief compared to standard care. Scores range from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores reflect worse pain intensity. This measure focuses on immediate postoperative pain change.
Change in Opioid Consumption for Postoperative Pain | 12 weeks (monitored throughout the study duration)
  Measure the amount of opioid medication administered for postoperative pain relief among patients in each group. This outcome evaluates whether the increase in TENS use changes the need for opioid pain management, contributing to safer postoperative care. Scores are measured in milligrams, where higher values reflect a worse outcome.
Change in Postoperative Discharge Time | Measured at discharge, within the first 12 weeks post-intervention
  Track the time from surgery to patient discharge in each group (Control, Education, and Nudging) to assess whether increased TENS use facilitates faster recovery. Shorter discharge times indicate improved postoperative recovery, likely linked to better pain management and decreased reliance on opioids. Scores are measured in minutes, where higher values reflect a worse outcome.

OTHER OUTCOMES:
Healthcare Staff Perceptions of Educational and Nudging Interventions | Collected after the final intervention phase (approximately 3 weeks)
  Conduct in-depth interviews with 20-25 anesthesia staff members to explore their experiences of the educational and nudging interventions aimed at increasing TENS usage. This outcome will provide insights into facilitators and barriers to TENS adoption, as well as the acceptability and perceived impact of behavioral interventions in a clinical setting.
Patient Experiences of TENS for Postoperative Pain Management | Collected within 1-2 days post-discharge
  Conduct interviews with 20-25 patients who underwent urological surgery and received TENS as part of their postoperative care. The interviews will explore patients' perspectives on pain relief, ease of TENS use, and the perceived impact on postoperative symptoms such as urinary urgency and bladder spasms. This outcome will help assess patient satisfaction and the subjective effectiveness of TENS in enhancing recovery.

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Sahlgrenska university hospital, Gothenburg, VGR
  - Sahlgrenska university hospital, Gotborg
  - Sahlgrenska University Hospital, Gothenburg
  - Sahlgrenska university hospital, Gothenburg